CLINICAL TRIAL: NCT05938907
Title: Effect of Concentrated Growth Factors on Healing of Apicomarginal Defects: a Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wen Luo, Associate Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RH2200003294
Record Dates: First submitted 2023-06-22; First posted 2023-07-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Concentrated Growth Factor; Bone Substitute
MeSH Terms: interventions — Bone Substitutes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- only apical surgery group (No Intervention): which will undergo only apical surgery (including apicoectomy, inflammation debridement, and retrofilling of the root apex)
- bone substitute group (Experimental): which will undergo apical surgery plus bone substitute
  Interventions: Other: bone substitute
- concentrated growth factors group (Experimental): which will undergo apical surgery plus CGF (concentrated growth factors)
  Interventions: Other: concentrated growth factor
- bone substitute and CGF group (Experimental): which will undergo apical surgery plus bone substitute and CGF gel
  Interventions: Combination Product: concentrated growth factor + bone substitute

INTERVENTIONS:
Other: concentrated growth factor — Implanting concentrated growth factor into the area of root apical bone defect
  Arms: concentrated growth factors group
Other: bone substitute — Implanting bone substitute into the area of root apical bone defect
  Arms: bone substitute group
Combination Product: concentrated growth factor + bone substitute — Implanting concentrated growth factor + bone substitute into the area of root apical bone defect
  Arms: bone substitute and CGF group

SUMMARY:
The persistent and chronic apical periodontitis has caused great difficulties for clinical physicians. Ensuring rapid and successful healing of the extensively damaged periapical region is a pressing issue that needs to be addressed. The treatment options include traditional apical surgery, simultaneous placement of bone powder and membrane after apical surgery, and simultaneous placement of sticky bone (bone powder mixed with concentrated growth factors gel) and membrane. However, high-quality evidence regarding these various treatment options is scarce. The purpose of this study is to compare the advantages and disadvantages of each treatment option, in order to guide clinical physicians in the application of apical surgery.

DETAILED DESCRIPTION:
This prospective study will recruit 72 patients with chronic periapical periodontitis in their anterior teeth or premolars, all of which have received comprehensive root canal treatment. The patients will be randomly divided into four groups: Group A, which will undergo only apical surgery (including apicoectomy, inflammation debridement, and retrofilling of the root apex); Group B, which will undergo apical surgery plus bone powder; Group C, which will undergo apical surgery plus CGF (concentrated growth factors); and Group D, which will undergo apical surgery plus bone powder and CGF gel. Each group will consist of 18 patients, and all surgeries will be performed by the same experienced doctor. The participants will receive a 1-year follow-up with the assistance of a professional doctor, including questionnaire data and daily records of pain and swelling at 2, 6, and 12 hours and 7 days after the intervention. Cone-beam computed tomography (CBCT) images will also be taken before the surgery, immediately after the surgery, and at 2, 3, 4, 6, and 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above.
* Tooth with significant symptoms or with root apex bone tissue destruction that cannot be treated by non-surgical methods.
* The affected tooth is either an anterior tooth or a premolar.
* The size of the lesion during preoperative cone beam computed tomography (CBCT) coronal acquisition is at least 6 mm but not more than 12 mm.
* The affected tooth has undergone successful root canal treatment.
* CBCT shows intact lingual side bone plate in the apical region, with only buccal alveolar bone defect present.
* Good oral hygiene and compliance with medical instructions.

Exclusion Criteria:

* Severe periodontal destruction, with over 1/3 of the root length absorbed by alveolar bone.
* CBCT shows root fracture or root canal perforation.
* After root apex surgery, crown-root ratio ≤1:1.
* Presence of surgical contraindications, systemic and local factors that affect wound healing.
* Pregnant women and females planning to conceive within the next two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Root apex healing status | up to 12 months
  Measurements of postoperative apical bone healing were obtained using cone-beam computed tomography (CBCT) in horizontal, coronal, and sagittal planes, respectively.
  Unit: mm

SECONDARY OUTCOMES:
pain status | 7 days
  Record the pain condition of patients postoperatively at 2, 6, and 12 hours, as well as daily for 7 days after the surgery through questionnaire surveys.
  The pain scale is as follows:
  0: No pain;
  1. (mild): Discomfort or pain that is felt but does not require medication;
  2. (moderate): Pain that is uncomfortable but tolerable, and can be effectively relieved with pain medication;
  3. (severe): Pain that is difficult to bear.
postoperative swelling | 7 days
  Record the postoperative swelling of patients postoperatively at 2, 6, and 12 hours, as well as daily for 7 days after the surgery through questionnaire surveys.
  Postoperative swelling score will be rated on the following scale:
  0: No swelling;
  1. Mild swelling at the surgical site;
  2. Moderate swelling outside the surgical area;
  3. Severe swelling outside the treatment area.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No